CLINICAL TRIAL: NCT05014620
Title: Exploring Caregiver Representations That Could be Obstacles or Elements Favouring the Implementation of a Therapeutic Education Programme for Mental Health Patients: a Multicentre Qualitative Study.
Acronym: ETPsy
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: RAT APPARA 2018
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Therapeutic Patient Education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-directive interview — semi-structured exploratory interview

SUMMARY:
Therapeutic patient education (TPE) is one of the approaches used to manage chronic diseases. It aims to make the patient an active participant in his or her own care and to establish an effective partnership with the carer, thereby also responding to the need to control health expenditures.

However, the contribution of TPE has revolutionised healthcare professions, in particular by profoundly changing the carer-patient relationship and certain aspects of their professional culture.

a recent action-research study conducted in partnership with Crf-Cnam in Paris showed that although the training of professionals appears to be a major issue, the integration of TPE forces the involved parties to question their practices. TPE imposes a change in the understanding that carers have of their usefulness in accompanying patients and in their perception of education and care. It also changes their relationship to the involvement of patients in maintaining their health.

The implementation of educational approaches in Mental Health is also at the origin of many questions.

In a study of patients suffering from schizophrenia, discrepancies appeared amongst the carers, whose outlooks seemed to be correlated with their experience in TPE. The carer-caregiver relationship was evoked with a feeling of lack of exchange, and a feeling of infantilization for certain carers. This study highlights the misconception that some psychiatric caregivers have of TPE in somatic care, and the idea that TPE is limited to drug treatments.

Therapeutic education is of particular importance as it is a determinant of the schizophrenic patient's adherence to therapeutic principles. However, it must be based on an appropriate strategy that facilitates communication and the exchange of knowledge with patients suffering from severe and persistent psychological disorders.

During the implementation of two ongoing TPE programs initiated with schizophrenic patients, we were able to observe that despite the knowledge of the TPE caregivers, there were still difficulties in its implementation: lack of recruitment, organizational difficulties, loss of motivation...

In the same prism as the development of new care strategies by the Ministère des solidarités et de la santé, we asked ourselves questions about strengthening the training of paramedical staff, such as: how can health literacy be enriched in mental health training programs? But the trainig of individuals in the field seems to be only one of the components. This care project raises questions about values systems and the mechanisms for legitimizing power, and requires consent and commitment from the various actors.

The hypothesis formulated is that one of the keys to better patient adherence and better appropriation of a TPE programme in mental health would be to take into account the representations of the carers dispensing these programmes. This investigation will be based on TPE programs dispensed to schizophrenic patients at La Chartreuse Psychiatric Hospital in Dijon, France.

ELIGIBILITY:
Inclusion Criteria:

* Person agreeing to participate;
* Paramedical and medical caregivers (nurses, head nurses, nursing assistants, dieticians, social workers, pharmacists, dentists, doctors) practicing in psychiatry;
* Dispensing / having dispensed in the past 12 months a TPE program ( among the following programs : "Quand la Psych...Ose" and/or "EBENE") for patients with schizophrenic disorders (Group 1 and 2) or having never provided a TPE program (Group 3).

Exclusion Criteria:

- Paramedical and medical caregivers who have already provided the two TPE programs listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical and paramedical staff providing a TPE program
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Characteristics of the representations of medical and paramedical caregivers providing or not providing a TPE program in Mental Health | Through study completion, an average of 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Rat C, Meunier-Beillard N, Moulard S, Denis F. Caregiver Representations of Therapeutic Patient Education Programmes for People with Schizophrenia: A Qualitative Study. Healthcare (Basel). 2022 Aug 29;10(9):1644. doi: 10.3390/healthcare10091644. PMID 36141256